CLINICAL TRIAL: NCT02577718
Title: Phase 1/2 Study to Evaluate the Safety and Effectiveness of Novel Non-Antibiotic, Non-Heparin Nitroglycerin Based Catheter Lock Solution Used for the Prevention of Intraluminal Central Venous Catheter (CVC) Infections in Cancer Patients
Brief Title: Safety and Effectiveness of Novel Nitroglycerin Based Catheter Lock Solution
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novel Anti-Infective Technologies, LLC (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NiCE
Record Dates: First submitted 2015-10-13; First posted 2015-10-16 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Catheter-Associated Infections; Catheter-Related Infections
MeSH Terms: conditions — Catheter-Related Infections

ARMS (1):
- Nitroglycerin-Citrate-Ethanol (NiCE) (Experimental): Antimicrobial Nitroglycerin-Citrate-Ethanol catheter lock solution was administered for 2 hours then flushed
  Interventions: Drug: Nitroglycerin-citrate-ethanol (NiCE)

INTERVENTIONS:
Drug: Nitroglycerin-citrate-ethanol (NiCE) — Lock solution instilled in catheter lumens for 2 hours then flushed. Administration for up to 30 days, daily as in-patient or once weekly as out-patient

SUMMARY:
The objective of this Phase I/II pilot study is to evaluate the safety and effectiveness of a non- antibiotic chelator based lock solution that contains nitroglycerin in combination with sodium citrate and ethanol (NiCE lock solution) for prevention of central line associated bloodstream infection (CLABSI).

* The primary objective of this study is to evaluate the safety and estimate the rate of adverse events associated with the NiCE lock solution.
* The second primary objective is to estimate the rate of CLABSI in patients receiving the NiCE lock solution.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients who have a long term central venous catheter (CVC)-and the CVC has been in place for at least 14 days and is expected to remain in place at least for 30 days after enrollment
* The CVC consists of a 5.0 French size, dual-lumen, peripherally inserted central catheter
* Patients who are willing and capable to provide Informed Consent
* Patients who are willing and capable to follow the instructions required to complete the study
* Females (of child bearing potential) and males (of child bearing potential) must be abstinent or agree to use birth control during the study.

Exclusion Criteria:

* Patients who have an antimicrobial CVC.
* Patients who have a short term CVC that have been placed in ICU (mainly rigid wall CVCs placed for acute care in ICU).
* Patients who are hypotensive with a systolic blood pressure reading of <110 mmHg at any time over the 3 days prior to study entry
* Patients who are not awake, not alert, or who cannot express pain or discomfort related to the catheter locks
* Patients with an existing local or systemic infection as defined by evidence of fever (a body temperature > 38.0o C with two readings taken at least 10 minutes apart or one body temperature > 38.3o) and any of the following within 24 hours of enrollment: Pulse rate > 100 beats/min.; Respiratory rate > 20/min.; WBC count >12,000/mm3, <4,000/mm3 or differential count showing >10% band forms. Patient will still be eligible for the study if the participant's white blood cell count (WBC) is outside normal limits due to chemotherapy treatment or underlying conditions. Systolic blood pressure <90 mm Hg.
* Signs and symptoms of localized catheter-related infection (tenderness and/or pain, erythema, swelling, purulent exudates within 2 cm of entry site)
* Patients with an occluded (partially or totally) catheter defined as inability to either withdraw blood or instill 3cc of fluid without resistance through any catheter lumen
* Patients with multiple co-existing central venous catheters at the time of enrollment will not be enrolled.
* Patients in whom the lock solution application will interfere with routine treatment of the underlying disease
* Patients with a known history of allergic reaction to ethanol, nitroglycerin, or citrate.
* Female patients who are pregnant or breast feeding
* Patients who are on disulfiram, metronidazole or are dependent on alcohol
* Patients receiving phosphodiesterase type 5 (PDE-5) inhibitors (such as sildenafil, tadalafil, vardenafil).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06-22 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Chaftari AM, Hachem R, Szvalb A, Taremi M, Granwehr B, Viola GM, Amin S, Assaf A, Numan Y, Shah P, Gasitashvili K, Natividad E, Jiang Y, Slack R, Reitzel R, Rosenblatt J, Mouhayar E, Raad I. A Novel Nonantibiotic Nitroglycerin-Based Catheter Lock Solution for Prevention of Intraluminal Central Venous Catheter Infections in Cancer Patients. Antimicrob Agents Chemother. 2017 Jun 27;61(7):e00091-17. doi: 10.1128/AAC.00091-17. Print 2017 Jul. PMID 28416559

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NiCE Lock
Started | 60
Completed | 52
Not Completed | 8
Not completed — Death | 6
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | NiCE Lock
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 67 [26 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 49
  More than one race | 0
  Unknown or Not Reported | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60
Number of patients with Hypertension [Count of Participants; unit: Participants] — Number
  Participants | 36
Type of Cancer [Count of Participants; unit: Participants]
  Acute Lymphatic Leukemia | 12
  Acute Monocytic Leukemia | 34
  Lymphoma | 1
  Aplastic Anemia | 1
  Myelofibrosis | 1
  Chronic Lymphatic Leukemia | 1
  Chronic Monocytic Leukemia | 3
  Acute Myelogenous Leukemia | 2
  Myelodysplastic Syndrome | 3
  B cell Acute Lymphatic Leukemia | 1
  Biphenotypic acute leukemia | 1
Median Standard Deviation of Systolic Blood Pressure [Median (Full Range); unit: mm Hg] | 7.86 [1.15 to 41.48]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Drug-Related Hypotension
Description: Drug-related hypotension is defined as a significant drop in measured blood pressure (BP) that exceeds the normal BP variability of a patient by 30%, that is associated with clinical signs and symptoms (dizziness and syncope) and is unexplained by factors other than the lock solution (such as other antihypertensive drugs, sepsis, bleeding). BP variability will be based on the standard deviation (SD) of a patient's blood pressure measured in the 3 days preceding participation in this trial and will be calculated at the time of trial entry.
Time Frame: From date of randomization until date of first Drug-Related Hypotension within 10 minutes of each flush, assessed up to 60 days
Population: All patients receiving at least one dose
Measure: Count of Participants; unit: Participants
Groups:
- NiCE Lock: All patients who received at least one dose
Arm/Group | NiCE Lock
Number analyzed (Participants) | 60
Participants | 0

2. Secondary Outcome: Incidence of Catheter-Associated Infections
Description: Catheter-Associated Infections will be measured by microbiological culture defined as either Catheter-Related Bloodstream Infection (CRBSI) as defined by the Infectious Diseases Society of America (IDSA), particularly in neutropenic patients, or Central Line-Associated Bloodstream Infection (CLABSI) as defined by the Centers for Disease Control and Prevention (CDC), particularly in non-neutropenic patients
Time Frame: 60 Days
Population: 619 catheter days on NiCE Lock Solution / 1853 catheter days off NiCE Lock Solution
Measure: Number; unit: infections per 1000 catheter days
Units Other Than Participants: catheter days
Groups:
- NiCE Lock: Days when patients received NiCE Lock
- Off NiCE Lock: Days patients did not receive NiCE Lock
Arm/Group | NiCE Lock | Off NiCE Lock
Number analyzed (Participants) | 60 | 60
Number analyzed (catheter days) | 619 | 1853
infections per 1000 catheter days | 0 | 1.6

ADVERSE EVENTS:
Groups:
- NiCE Lock: Patients had days they received NiCE Lock and days they did not receive NiCE Lock (off-Lock days). NiCE Lock was a combination of three different agents so combined results are presented. Most patients received NiCE Lock with Nitroglycerin 30 μg/ml.
Arm/Group | NiCE Lock
All-Cause Mortality (participants affected / at risk) | 6/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 2/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NiCE Lock (N=60)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — Transient Rash, occurred after 23rd dose, resolved
Headache (transient) (Nervous system disorders) | 1 (1) — Mild, Transient Headache reported after 4th of 5 doses, resolved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No